CLINICAL TRIAL: NCT07337980
Title: A Study on the Safety and Effectiveness of Endoscopic Intracavitary Submucosal Dissection for Gastric Extracavitary-Type Submucosal Tumors
Status: Not yet recruiting | Type: Observational
Sponsor: Zhongda Hospital (Other)
Responsible Party: Principal Investigator, Ruihua Shi, Professor, Zhongda Hospital
Other Study IDs: GI of Zhongda Hospital
Record Dates: First submitted 2026-01-03; First posted 2026-01-13 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Interstitialoma; Endoscopic Surgery
Keywords: endoscopic surgery; interstitialoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Endoscopic-surgery Group: Patients with extraluminal growing stromal tumors undergoing endoscopic treatment
  Interventions: Procedure: Extraluminal growing stromal tumors treated endoscopically

INTERVENTIONS:
Procedure: Extraluminal growing stromal tumors treated endoscopically — To observe the safety and efficacy of endoscopic treatment of extraluminal growing stromal tumors

SUMMARY:
The aim of this study is to explore the safety and efficacy of endoscopic surgery in the treatment of extraluminal growing stromal tumors

DETAILED DESCRIPTION:
The aim of this study is to explore the safety and efficacy of endoscopic surgery in the treatment of extraluminal growing stromal tumors

ELIGIBILITY:
Inclusion Criteria:

* (1) CT scan showed extramural protrusion of the stomach (2) ultrasonic endoscopy revealed submucosal tumors with extra-gastric growth; (3) patients received ESD/EFTR or surgical treatment

Exclusion Criteria:

* (1) patients had malignant tumors in the stomach or had undergone stomach surgery (2) follow-up records were incomplete.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with gastric stromal tumor with extraluminal growth
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2026-12-12 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Complete resection rate | 12 months
  Complete resection rate of extraluminal growing stromal tumors

SECONDARY OUTCOMES:
Recurrence-free survival | 12 months
  Recurrence-free survival of extraluminal growing stromal tumors after surgery

IPD SHARING:
Plan to Share IPD: Undecided
Since this data may involve the privacy of patients, hospital ethics should be followed.